CLINICAL TRIAL: NCT06051968
Title: Effects of an Online Hearing Rehabilitation Support for First-time Hearing Aid Users: A Randomised Controlled Trial.
Brief Title: Effects of an Online Hearing Support for First-time Hearing Aid Users
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Horselvarden Region Ostergotland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-01633-02
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Hearing Loss; Hearing Impairment; Hearing Disorders; Hearing Disability; Ear Diseases; Sensation Disorders; Otorhinolaryngologic Diseases
MeSH Terms: conditions — Hearing Loss; Hearing Disorders; Ear Diseases; Sensation Disorders; Otorhinolaryngologic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants get hearing rehabilitation according to common practice and the online hearing support.
  Interventions: Behavioral: Online hearing support for first-time hearing aid users
- Control group (Active Comparator): Participants get hearing rehabilitation according to common practice.
  Interventions: Behavioral: Hearing rehabilitation according to common practice.

INTERVENTIONS:
Behavioral: Online hearing support for first-time hearing aid users — Participants get hearing rehabilitation according to common practice and the online hearing support consists of five chapters that aim to give information, support, and advice to the new hearing aid users. The participants are assigned a new chapter between each visit at the clinic.
  Other Names: Stöd och Behandling för nya hörapparatanvändare; Internetbaserat stöd vid hörselrehabilitering
  Arms: Intervention group
Behavioral: Hearing rehabilitation according to common practice. — Participants get hearing rehabilitation according to common practice.
  Arms: Control group

SUMMARY:
The goal of this randomised controlled trial is to test a online hearing support for first-time hearing aid users. The main questions it aims to answer are short- and long-term effects on the emotional and social consequences of hearing loss that the participants experience, use of communications strategies, experienced listening in complex sound environments and perceived effectiveness and satisfaction with hearing aids.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 20 years of age that are eligible for hearing aids
* Access to a computer, tablet and/or smartphone with internet
* Access to a Swedish BankID or equivalent

Exclusion Criteria:

* Inability to read and understand Swedish

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The Hearing Handicap Inventory for the Elderly (HHIE) | Baseline, directly post intervention and 6 months post intervention.
  Assessing changes in emotional and social effects of hearing loss, self-perceived activity limitations and participation restrictions. Minimum 0 points to maximum 100 points. Higher score indicates greater emotional and social effects of hearing loss.

SECONDARY OUTCOMES:
The 12-item Speech, Spatial and Qualities of Hearing Scale (SSQ12) | Baseline, directly post intervention and 6 months post intervention.
  Assessing experience of listening in complex sound environments. Minimum 0 points to 120 points. Higher score indicates less problems with hearing in the specified situations.
Communication Strategies Scale (CSS) | Baseline, directly post intervention and 6 months post intervention.
  Assessing changes in use of verbal, non-verbal and maladaptive communication strategies. Minimum 25 points to maximum 125 points. Higher score indicates a greater use of communication strategies.
The International Outcome Inventory for Hearing Aids (IOI-HA) | Directly post intervention and 6 months post intervention.
  Assessing changes in perceived effectiveness and satisfaction with hearing aids.
  Minimum 7 points to maximum 35 points. Higher score indicates higher perceived effect.

OTHER OUTCOMES:
Subjective impact of the intervention, reported by the users: Memory of the intervention | 6 months post intervention
  The participants are asked what they remember from their intervention.
Subjective impact of the intervention, reported by the users: Seeking more or other information | 6 months post intervention
  The participants are asked if they searched for more or other information about hearing or hearing aids.
Subjective impact of the intervention, reported by the users: Adverse effects | 6 months post intervention
  The participants are asked if they experienced any adverse effects of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Öberg, Principal Investigator — Horselvarden Region Ostergotland
Locations (1):
- Audiologimottagningen Lund, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No